CLINICAL TRIAL: NCT07339774
Title: Chinese Herbal Oral Solution and Mouthwash Shorten the Duration of Severe Radiotherapy-induced Oral Mucositis in Patients With Head and Neck Malignancies.
Brief Title: Traditional Chinese Medicine Preparation Alleviates Radiotherapy-induced Oral Mucositis in Head and Neck Cancer Patients.
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Xingchen Peng, Ph.D, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024(1774)
Record Dates: First submitted 2025-12-02; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Radiotherapy-induced Oral Mucositis
MeSH Terms: interventions — Mouthwashes; Radiotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zishui Daohuo oral liquid combined with Kujiu mouthwash group. (Experimental)
  Interventions: Drug: Zishui Daohuo oral liquid combined with Kujiu mouthwash; Radiation: Radiotherapy
- Placebo oral liquid and mouthwash (Placebo Comparator)
  Interventions: Drug: Placebo oral liquid and mouthwash; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Placebo oral liquid and mouthwash — Placebo oral liquid and mouthwash with the same color, aroma, and taste as the experimental group, and without any related drug ingredients
  Arms: Placebo oral liquid and mouthwash
Drug: Zishui Daohuo oral liquid combined with Kujiu mouthwash — Oral administration of Zishui Daohuo oral liquid combined with gargling using Kujiu mouthwash.
  Arms: Zishui Daohuo oral liquid combined with Kujiu mouthwash group.
Radiation: Radiotherapy — One of the inclusion criteria for the study was that patients with squamous carcinoma of the head and neck (including nasopharyngeal carcinoma) needed to receive either radiotherapy alone or simultaneous radiotherapy and chemotherapy.

SUMMARY:
Evaluate the effectiveness and safety of traditional Chinese medicine compound in improving radiotherapy-induced oral mucositis in patients with head and neck malignant tumors.

DETAILED DESCRIPTION:
The aim of this clinical trial is to evaluate the efficacy and safety of combining a traditional Chinese medicine (TCM) oral solution with a mouthwash in reducing the duration of severe radiation-induced oral mucositis (RIOM). The study addresses two primary questions: (1) whether the combined use of the TCM oral solution and mouthwash can effectively shorten the duration of severe RIOM, and (2) whether their use is associated with adverse events in patients undergoing radiotherapy.

Participants will initiate treatment on the first day they develop severe RIOM (RTOG grade ≥3) during radiotherapy. They will take Zishui Daohuo oral solution three times daily and use Kuju gargling solution six times daily, or matched placebos. Treatment will continue until two weeks after completion of radiotherapy. After each administration, patients must refrain from eating, drinking, or performing oral hygiene for at least one hour to maximize mucosal contact time.

The trial will compare the intervention group with the placebo group to determine the potential benefits of the combined regimen in improving RIOM.

ELIGIBILITY:
Inclusion Criteria:

1. Patients pathologically diagnosed with non-metastatic head and neck malignant tumors;
2. Age range: 18 to 65 years old (including 18 and 65 years old);
3. Eastern Cooperative Oncology Group performance status of ≤2;
4. Radiotherapy or concurrent chemoradiotherapy is required;
5. The main organ functions well;
6. Sign informed consent.

Exclusion Criteria:

1. Allergic constitution (such as those known to be allergic to two or more drugs);
2. Patients who plan to use drugs that can cause or worsen oral mucosal inflammation (such as anti EGFR monoclonal antibodies, immune checkpoint inhibitors, etc.) after the start of radiotherapy;
3. Use of antibiotics, antifungal drugs, or antimicrobial mouthwash within 1 month of the study;
4. Poor oral hygiene and/or severe periodontal diseases;
5. History of head and neck radiotherapy;
6. Deemed unsuitable for the study by the investigators (concomitant with any other severe diseases).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
The duration of severe oral mucositis (RTOG grade≥3) | From the start of radiotherapy to 8 weeks after completion of radiotherapy.The evaluation period is approximately 14 weeks and 14.5 weeks.
  The Radiation Therapy Oncology Group (RTOG) toxicity criteria were utilized to assess RIOM. Grade 0 shows no change from baseline; Grade 1 of RIOM is associated with mucosal erythema or hyperemiam,and may cause mild pain not requiring analgesics. Grade 2 presents with patchy mucositis that may produce an inflammatory serosanguinous discharge and may be associated with moderate pain; Grade 3 consists of confluent, fibrinous mucositis and may include severe pain requiring narcotics; Grade 4 is characterized by ulceration, hemorrhage, or necrosis. Grades 1 and 2 are considered mild to moderate, while grades 3 and 4 are classified as severe.

SECONDARY OUTCOMES:
The time to onset of severe oral mucositis (RTOG grade≥3) | From the start of radiotherapy to 8 weeks after completion of radiotherapy.The evaluation period is approximately 14 weeks and 14.5 weeks.
  Time from the first day of radiotherapy to the first determination of SOM.
The duration of any-grade oral mucositis (OM) | From the start of radiotherapy to 8 weeks after completion of radiotherapy.The evaluation period is approximately 14 weeks and 14.5 weeks.
  The first determination of OM to the first instance of non-OM, without a subsequent instance of OM.
The time to onset of any-grade oral mucositis (OM) | From the start of radiotherapy to 8 weeks after completion of radiotherapy.The evaluation period is approximately 14 weeks and 14.5 weeks.
  Time from the first day of radiotherapy to the first determination of OM.
Relief rate of oral mucositis | From the start of radiotherapy to 8 weeks after completion of radiotherapy.The evaluation period is approximately 14 weeks and 14.5 weeks.
  The proportion of patients whose oral mucositis resolved to RTOG grade 0 at 4 and 8 weeks after completion of radiotherapy.
Adverse events | From the first day of radiotherapy to the day of the last radiation dose received, usually 6 or 6.5 weeks.
  Common Terminology Criteria for Adverse Events (CTCAE) 5.0 version

OTHER OUTCOMES:
The longitudinal dynamics of salivary microbiota | 1 week before radiotherapy, the middle of radiotherapy (3 weeks after the start of radiotherapy), and the end of radiotherapy (the last radiation dose received, usually 6 or 6.5 weeks).
  Unstimulated whole saliva samples will be collected via spitting method at three time points: baseline, mid-term radiotherapy (the week corresponding to 50% completion of the planned radiation fractions), and the end of radiotherapy (the final week of RT). 16S rRNA gene sequencing will be performed to assess alterations in the oral microbiota.
Analysis of Inflammatory Indicators in Oral Saliva | The time period is the period from the start of radiotherapy to the completion of radiotherapy.The evaluation period is approximately 6 weeks and 6.5 weeks.
  Measurement of circulating levels of interleukin-1β (IL-1β), interleukin-6 (IL-6), and tumor necrosis factor-alpha (TNF-α) in patient oral saliva.
Oral activities scores | The time period is the period from the start of radiotherapy to the completion of radiotherapy. The evaluation period is approximately 6 weeks and 6.5 weeks.
  Patients report the degree to the impact of MTS on oral activities (including swallowing, drinking, eating, talking, sleeping) (Likert scale 1 to 5) via the oral mucositis weekly questionnaire (OMWQ). Higher score indicates more severe symptoms.
TCM syndrome score for RIOM | From the start of radiotherapy to 8 weeks after completion of radiotherapy.The evaluation period is approximately 14 weeks and 14.5 weeks.
  The Radiation-Induced Oral Mucositis Symptom Score Scale is a 17-item patient-reported outcome measure assessing the severity of radiotherapy-related oral mucositis symptoms. The scale covers both oral local manifestations and systemic discomforts. Each item is rated on a 4-point Likert scale (0-3) corresponding to no, mild, moderate, and severe symptoms, respectively. The total score is calculated by summing the scores of all items. Higher total scores indicate greater symptom severity and a heavier symptom burden, whereas lower scores reflect milder symptoms or better symptom relief.
Mouth and throat soreness (MTS) scores | The time period is the period from the start of radiotherapy to the completion of radiotherapy.The evaluation period is approximately 6 weeks and 6.5 weeks.
  Patients report mouth and throat soreness (MTS) scores (Likert scale 1 to 5) via the oral mucositis weekly questionnaire (OMWQ). Higher score indicates more severe symptoms
Overall Health Status and Core Dimensions of Quality of Life | From the start of radiotherapy (baseline) to 2 months after treatment completion. The total evaluation period is approximately 14 to 14.5 weeks.
  European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) This instrument is a 30-item patient-reported outcome (PRO) measure designed to evaluate core aspects of health-related quality of life in cancer patients, including 5 functional scales (physical, role, cognitive, emotional, social), 3 symptom scales (fatigue, pain, nausea and vomiting), one global health status/quality of life scale, and 6 single-item symptom measures. Scores are linearly transformed to a range of 0-100. For the functional scales and the global health status scale, higher scores indicate better functional levels or quality of life; for the symptom scales/items, higher scores indicate greater symptom burden.
Head and Neck Cancer-Specific Symptoms | From the start of radiotherapy (baseline) to 2 months after treatment completion. The total evaluation period is approximately 14 to 14.5 weeks.
  The EORTC QLQ-H&N35 is a patient-reported outcome (PRO) instrument specifically designed to assess disease-related symptoms and treatment-related side effects in patients with head and neck cancer. It comprises 35 items, organized into seven multi-item subscales (pain, swallowing, senses, speech, social eating, social contact, and sexuality) and eleven single-item measures (such as dental problems, problems opening mouth, sticky saliva, coughing, etc.). All subscale and single-item scores are linearly transformed to a 0-100 scale using a standardized scoring algorithm. Interpretation of Scores: For all subscales and single items, higher scores represent more severe symptoms or greater symptom burden.
Xerostomia | 1 week before radiotherapy ; at the middle of radiotherapy (3 weeks after the start of radiotherapy) ; at the end of radiotherapy (the last radiation dose received, usually 6 or 6.5 weeks); and 1, 3 months after the end of radiotherapy.
  Xerostomia was graded per CTCAE v5.0 (Grade 1-4), with higher grades indicating worse symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Xingchen Peng, Professor, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Chengdu, Sichuan, China